CLINICAL TRIAL: NCT04122846
Title: Internet-based Emotional Awareness and Expression Therapy for Somatic Symptom Disorder
Acronym: MBS1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Stockholm University (Other)
Responsible Party: Principal Investigator, Robert Johansson, Associate professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KIMBS1
Record Dates: First submitted 2019-10-04; First posted 2019-10-10 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Somatic Symptom Disorder

STUDY DESIGN:
Intervention Model Description: Emotional Awareness and Expression Therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Emotional Awareness and Expression Therapy) (Experimental): Internet-based Emotional Awareness and Expression Therapy
  Interventions: Behavioral: Emotional Awareness and Expression Therapy

INTERVENTIONS:
Behavioral: Emotional Awareness and Expression Therapy — Very much based on "Unlearn your pain" by Howard Schubiner.

SUMMARY:
The main purpose of the study is to conduct an initial feasibility evaluation of the new Internet-based EAET treatment manual. We will include 50 patients with somatic symptom disorder to take part of the treatment for nine weeks through the Internet. A within-subject design will be used. Self-report measures of symptom level and mechanisms of change will be conducted weekly. Feedback on content, process and potential caveats will be collected using surveys and written evaluations from the participants at post-treatment. Linear mixed models will be used to investigate trajectories of change in symptoms and processes.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* A total score ≥10 on the PHQ-15
* A diagnosis of SSD according to the DSM-5, i.e ≥1 of the 3 of: disproportionate thoughts about the somatic symtom, persistently high level of anxiety, or excessive time and energy devoted in regard to symptoms or health concerns
* Symptom duration ≥6 months
* Written statement from a medical professional that states that a medical evaluation has been conducted.

Exclusion Criteria:

* Alcohol or substance addiction
* A diagnosis of a psychological condition that might require other treatment (e.g., psychosis, suicidality, etc)
* Other severe medical condition that might require other treatment
* Ongoing psychological intervention or psychotherapy that may interfere with the psychological treatment
* Ongoing medical treatment that may interfere with the psychological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
PHQ-15 | Baseline
  Patient Health Questionnaire Physical Symptoms
PHQ-15 | Weekly during treatment, for 9 weeks
  Change in physical symptoms (as measured by the PHQ-15)
PHQ-15 | At study completion, after 9 weeks
  Patient Health Questionnaire Physical Symptoms
PHQ-15 | At study completion, after 4 months
  Patient Health Questionnaire Physical Symptoms

SECONDARY OUTCOMES:
PHQ-9 | Baseline
  Patient Health Questionnaire Depression
PHQ-9 | At study completion, after 9 weeks
  Patient Health Questionnaire Depression
PHQ-9 | At study completion, after 4 months
  Patient Health Questionnaire Depression
GAD-7 | Baseline
  Patient Health Questionnaire Anxiety
GAD-7 | At study completion, after 9 weeks
  Patient Health Questionnaire Anxiety
GAD-7 | At study completion, after 4 months
  Patient Health Questionnaire Anxiety
SDS | Baseline
  Sheehan Disability Scale
SDS | At study completion, after 9 weeks
  Sheehan Disability Scale
SDS | At study completion, after 4 months
  Sheehan Disability Scale

OTHER OUTCOMES:
EPS-25 | Baseline
  Emotional Processing Scale (Measure of treatment process)
EPS-25 | Weekly during treatment, for 9 weeks
  Emotional Processing Scale (Measure of treatment process)
EPS-25 | At study completion, after 9 weeks
  Emotional Processing Scale (Measure of treatment process)
EPS-25 | At study completion, after 4 months
  Emotional Processing Scale (Measure of treatment process)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Johansson, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maroti D, Ek J, Widlund RM, Schubiner H, Lumley MA, Lilliengren P, Bileviciute-Ljungar I, Ljotsson B, Johansson R. Internet-Administered Emotional Awareness and Expression Therapy for Somatic Symptom Disorder With Centralized Symptoms: A Preliminary Efficacy Trial. Front Psychiatry. 2021 Feb 12;12:620359. doi: 10.3389/fpsyt.2021.620359. eCollection 2021. PMID 33679478